CLINICAL TRIAL: NCT03224845
Title: Transgenerational Prevention of Anxiety in Children at Ultra-high Risk
Brief Title: Courageous Parents, Courageous Children
Acronym: COACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1022588
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioural skills training (Experimental)
  Interventions: Behavioral: Cognitive behavioural skills training
- No intervention (No Intervention): Participants in the control group will receive their usual clinical care and will not be discouraged from seeking any intervention.

INTERVENTIONS:
Behavioral: Cognitive behavioural skills training — The intervention will be delivered in two stages: First, the parent with an anxiety disorder will attend between six and sixteen weekly sessions of cognitive behavioural skills training focusing on their own anxiety. They will work on developing behaviours that will help them become less anxious in the long-run and on learning to evaluate danger in a realistic way. Next, the parent will take part in four to eight weekly sessions of anti-anxiety parenting skills training aiming to help them transfer the skills that they learned into parenting their children. In the parenting intervention, the parents will be guided to gradually expose their children to new situations, build communication skills and confidence, in addition to general parenting skills and principles.
  Arms: Cognitive behavioural skills training

SUMMARY:
Anxiety disorders usually start in childhood and adolescence and are associated with social and occupational difficulties in adulthood. Children who have a parent with an anxiety disorder and who find new situations distressing and avoid them are at an increased risk for developing an anxiety disorder. Research suggests that anti-anxiety parenting can help children grow up courageous and calm. It is, however, difficult to parent in an anti-anxiety way when the parent has an anxiety disorder himself or herself.

This research study will test the efficacy of a new program designed to prevent the onset or persistence of anxiety disorders in children at risk for anxiety disorders. The investigators will first help parents learn skills to cope with their own anxiety and then coach them to share these skills with their children and parent in an anti-anxiety way. The goal is to intervene early enough in the children's lives so that they can be free of anxiety disorders and lead happy, healthy and productive lives in adulthood.

ELIGIBILITY:
Parents:

Inclusion criteria:

Parents will be included if they have a current diagnosis of at least one anxiety disorder, one or more children between the ages two and eight years in their own care, capacity to provide informed consent, and ability to speak English well enough to benefit from the intervention.

Exclusion criteria:

Exclusion criteria for parents are receipt of an adequate course (6 or more sessions) of structured psychological therapy in the past 12 months, or plans to move out of Nova Scotia within the next three years. We will include parents with co-morbid mood disorders. However, those whose mood disorder is the primary complaint will be referred for treatment for their mood before being re-assessed. We will exclude parents with disorders that would interfere with the standard treatment protocol delivery; these include lifetime schizophrenia, autism, intellectual disability and current drug and alcohol use disorder.

Offspring:

Inclusion criteria:

Children are eligible if they are aged two to eight and if they have a score of inhibited temperament (negative emotionality) one standard deviation or more above the mean of an age-matched normative sample on the Laboratory Assessment of Temperament.

Exclusion criteria:

Those with lifetime schizophrenia, autism, general intellectual disability, and current drug and alcohol addiction will be excluded, as these conditions would impact on the standard delivery of the parenting intervention. We will exclude children currently receiving treatment for anxiety.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2017-09-17 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) | One year post randomization
  Diagnosis of anxiety disorder in the offspring
Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) | Two years post randomization
  Diagnosis of anxiety disorder in the offspring
Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) | Three years post randomization
  Diagnosis of anxiety disorder in the offspring
Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) | Five years post randomization
  Diagnosis of anxiety disorder in the offspring
Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) | Seven years post randomization
  Diagnosis of anxiety disorder in the offspring
Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) | Ten years post randomization
  Diagnosis of anxiety disorder in the offspring

SECONDARY OUTCOMES:
Teaching Task Battery | One year post randomization
  Parenting behaviours
Teaching Task Battery | Two years post randomization
  Parenting behaviours
Structured Clinical Interview for DSM-5 diagnoses (SCID-5) | One year post randomization
  Diagnosis of anxiety disorder in the parent
Structured Clinical Interview for DSM-5 diagnoses (SCID-5) | Two years post randomization
  Diagnosis of anxiety disorder in the parent
Laboratory Temperament Assessment Battery | One year post randomization
  Temperament in the offspring
Laboratory Temperament Assessment Battery | Two years post randomization
  Temperament in the offspring
Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) | Three years post randomization
  Diagnosis of major mood and psychotic disorders in offspring
Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) | Five years post randomization
  Diagnosis of major mood and psychotic disorders in offspring
Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) | Seven years post randomization
  Diagnosis of major mood and psychotic disorders in offspring
Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) | Ten years post randomization
  Diagnosis of major mood and psychotic disorders in offspring
Global Assessment of Functioning | One year post randomization
  Functioning in the offspring
Global Assessment of Functioning | Two years post randomization
  Functioning in the offspring
Global Assessment of Functioning | Three years post randomization
  Functioning in the offspring
Global Assessment of Functioning | Five years post randomization
  Functioning in the offspring
Global Assessment of Functioning | Seven years post randomization
  Functioning in the offspring
Global Assessment of Functioning | Ten years post randomization
  Functioning in the offspring
Screen for Child Anxiety Related Disorders | One year post randomization
  Anxiety in the offspring - continuous
Screen for Child Anxiety Related Disorders | Two years post randomization
  Anxiety in the offspring - continuous
Screen for Child Anxiety Related Disorders | Three years post randomization
  Anxiety in the offspring - continuous
Screen for Child Anxiety Related Disorders | Five years post randomization
  Anxiety in the offspring - continuous
Screen for Child Anxiety Related Disorders | Seven years post randomization
  Anxiety in the offspring - continuous
Screen for Child Anxiety Related Disorders | Ten years post randomization
  Anxiety in the offspring - continuous
Spence Children's Anxiety Scale | One year post randomization
  Anxiety in the offspring - continuous
Spence Children's Anxiety Scale | Two years randomization
  Anxiety in the offspring - continuous
Spence Children's Anxiety Scale | Three years post randomization
  Anxiety in the offspring - continuous
Spence Children's Anxiety Scale | Five years post randomization
  Anxiety in the offspring - continuous

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No